CLINICAL TRIAL: NCT01543672
Title: VOLUMES Treatment of Larger Tumor Volumes or ≥ 2 Lung Tumors Simultaneously in Lung Cancer Patients Using SBRT in a Mean-lung Dose Escalation Study
Brief Title: Irradiation of Large Lung Tumors or Two or More Lung Metastases Simultaneously
Acronym: VOLUMES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11VOL
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer; Metastatic Lung Cancer
Keywords: lung; SBRT; MLD; toxicity
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT group A (Experimental): escalate MLD in medically inoperable patients with tumors larger than 5 cm in diameter (primary or solitary metastases)
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- SBRT group B (Experimental): Escalate the MLD in patients with ≥ 2 lung metastases
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — 3-5 fractions within 10-14 days
  Other Names: Stereotactic Body Radiotherapy
  Arms: SBRT group A
Radiation: Stereotactic Body Radiotherapy (SBRT) — 3-5 fractions per tumor within one treatment session or sequential within one month
  Other Names: Stereotactic Body Radiotherapy
  Arms: SBRT group B

SUMMARY:
Treatment of larger tumor volumes or ≥ 2 lung metastases simultaneously in lung cancer patient using Stereotactic Body Radiation Therapy (SBRT) in a mean-lung dose escalation study.

DETAILED DESCRIPTION:
A phase I/II multicenter trial will be conducted in patients with medically inoperable with peripheral non small cell lung cancer (NSCLC) > 5 cm without lymph node involvement (group A) or medically with ≥ 2 or more lung metastases (group B). Radiation pneumonitis is expected to be dose-limiting in these patients and there is evidence that the incidence is predicted by the mean lung dose (MLD). The MLD escalation will be performed separately in both patient groups, using a time-to-event continual reassessment method (TITE-CRM). All patients will receive 3-5 fractions SBRT to the lung tumor(s), with a minimum mean PTV dose ≥ 42 Gy. Fraction size may be downscaled based on the MLD constraint.

ELIGIBILITY:
Inclusion Criteria for group A and B:

* Weight loss < 10% in the last three months.
* WHO-performance status ≤ 2
* Medical inoperable patients or patients refusing surgery.
* Chemotherapy is allowed in neoadjuvant and adjuvant setting, with exclusion of the period 4 weeks pre-SBRT and 6 weeks post-SBRT.
* Before patient registration, written informed consent must be given according to ICH/GCP, national and local regulations.

Risk group A specification:

* NSCLC (Cytological or histological proven) patients with peripheral tumors >5 cm with tumor staging cT2bN0M0 or cT3N0M0 (chest wall infiltration is no exclusion criteria, as long as the tumor diameter is > 5 cm).
* Single peripheral lung metastasis in inoperable patients with a diameter of > 5 cm. In case of first presentation of metastatic disease, cytological or histological proof is obligated.
* In patients without cytological or histological confirmation of NSCLC, a growing FDG-PET positive lesion (SUV >5) is accepted if a contra-indication for invasive diagnostic examination (or refusal) is present.

Risk group B specification:

* Patients with ≥ 2 simultaneous peripheral lung metastases ≤ 5 cm of any origin at any location in the lung.
* In case of first presentation of metastatic disease, cytological or histological proof is obligated. This is not necessary in case of a history of an already proven disseminated disease.
* Patients having ≥ 2 peripheral lung metastases without unacceptable dose overlap.

Exclusion Criteria:

* Patients with central tumors
* Pancoast tumors
* Prior radiotherapy treatment to the thorax
* Patients receiving any systemic treatment during SBRT
* Pregnant patients
* Patients previously treated with adriamycin agents in case of heart involvement within the treatment field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
MLD | 4 years
  The assessment of the maximum mean lung dose that can be safely treated with SBRT and that is associated with a 20% probability of the DLT.

SECONDARY OUTCOMES:
loco-regional control | 4 years
  Determine the local control and regional control as a function of the mean lung dose, the largest toxicity effects as a function of the MLD and the overall survival.
overall survival | 5 years
  Determine the local control and regional control as a function of the mean lung dose, the largest toxicity effects as a function of the MLD and the overall survival.
Quality of life assessment | 2 years
  valuate the increase or decrease of physical discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Peulen, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (5):
- United States (2):
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Thomas Jefferson University/ Kimmel Cancer Center, Philadelphia, Pennsylvania
- Prinses Margaret Hospital, Toronto, Ontario, Canada
- Universitätsklinikum Würzburg, Würzburg, Bavaria, Germany
- NKI-AVL, Amsterdam, Netherlands